CLINICAL TRIAL: NCT04086719
Title: An Open-Label, Single Sequence, Crossover Study to Investigate the Effects of OCT1 Inhibition Utilizing Pyrimethamine on Pharmacokinetics of BMS-986165 in Healthy Male Volunteers.
Brief Title: An Investigational Study to Determine the Drug Level Profile of BMS-986165 in Healthy Male Volunteers Following Transporter Inhibition.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM011-100
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — deucravacitinib; Pyrimethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS- 986185 + Pyrimethamine (Experimental)
  Interventions: Drug: Pyrimethamine
- BMS-986185 (Experimental)
  Interventions: Drug: BMS-986165

INTERVENTIONS:
Drug: BMS-986165 — Oral administration of tablet BMS- 986165
  Arms: BMS-986185
Drug: Pyrimethamine — Oral administration of Pyrimethamine in combination with BMS-986185
  Arms: BMS- 986185 + Pyrimethamine

SUMMARY:
Study of what the body does to drug BMS-986165 when it is taken together with pyrimethamine

ELIGIBILITY:
Inclusion Criteria:

* Patients must be willing and able to complete all study-specific procedures and visits
* Healthy patients, as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiogram, and clinical laboratory determinations
* Body mass index (BMI) of 18 to 32 kg/m2, inclusive, at screening
* Normal renal function at screening

Exclusion Criteria:

* Any medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of or active liver disease
* Current or recent (within 3 months of study drug administration) gastrointestinal disease that could impact upon the absorption of study drug
* History or presence of clinically significant acute or chronic bacterial, fungal, or viral infection (eg, pneumonia, septicemia) within the 3 months prior to screening
* Additional criteria may apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum comcentration (Cmax) | Day 1, Day 5
Area under the concentration-time curve from time zero extrapolated to AUC(INF) | Day 1, Day 5

SECONDARY OUTCOMES:
Incidences of Adverse Events (AE's) | Approximetly 20 days
Time of maximum observed concentration (Tmax) | Approxmiately 20 days
Half- life time (T-Half) | Day 1, Day 5
Apparent oral clearance (CL/F) | Day 5
Apparent volume of distribution at terminal phase (Vz/F) | Day 5
Ratio of metabolite AUC(0-T) to parent AUC(0-T) corrected for Molecular weight MRAUC(0-T) | Day 5
Ratio of metabolite AUC(INF) to parent AUC(INF) corrected for Moecular weight MRAUC(INF) | Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences - Salt Lake, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm